CLINICAL TRIAL: NCT07363785
Title: The Effects Of Therapeutic Touch Applied To Premature Infants On Behavioural Responses, Comfort And Physiological Parameters: A Randomised Controlled Trial
Brief Title: Therapeutic Touch in Premature Infants
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Habibe BAY, associate professor, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025/1144
Record Dates: First submitted 2026-01-06; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Premature Infants
Keywords: Preterm Infant; Therapeutic Touch; Behavioral Responses; Neonatal Comfort; Physiological Parameters
MeSH Terms: conditions — Premature Birth | interventions — Therapeutic Touch

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapeutic Touch group (Experimental): The babies in the intervention group will receive therapeutic touch twice a day, morning and evening, for one minute each time, for five days.
  Interventions: Behavioral: Therapeutic Touch
- Routine care group (No Intervention): Infants in the control group will continue with their routine clinical treatment and care without any intervention.

INTERVENTIONS:
Behavioral: Therapeutic Touch — Therapeutic Touch will be administered by the researcher to preterm infants in the intervention group under controlled environmental conditions. The care environment will be quiet, warm, and free from distracting stimuli, and infants will be positioned in a supine position for safe observation. The intervention will consist of gentle, stable, and rhythmic hand contact applied to the head, trunk, arms, and legs to promote relaxation and comfort. Therapeutic Touch will be applied twice daily for five consecutive days, with each session lasting approximately one minute. During the intervention, heart rate, respiratory rate, and oxygen saturation will be continuously monitored. Infants in the control group will receive routine neonatal care only.
  Arms: Therapeutic Touch group

SUMMARY:
Preterm birth is associated with increased physiological instability, stress responses, and developmental vulnerability due to immature organ systems and prolonged exposure to invasive procedures and environmental stressors in neonatal intensive care units (NICUs). In recent years, non-pharmacological, touch-based interventions have gained attention for their potential to support neurodevelopment, improve comfort, and stabilize physiological parameters in preterm infants.

Therapeutic Touch (TT) is a non-invasive, holistic intervention based on the modulation of the human energy field through gentle hand movements, aiming to reduce stress, promote relaxation, and support physiological regulation. Although TT has demonstrated beneficial effects in various populations, evidence regarding its effects on preterm infants remains limited.

This randomized controlled study aims to evaluate the effects of Therapeutic Touch on behavioral responses, comfort levels, and physiological parameters (heart rate, respiratory rate, oxygen saturation, and body temperature) in preterm infants hospitalized in the NICU. The findings are expected to contribute evidence for safe, supportive, and holistic neonatal care practices.

DETAILED DESCRIPTION:
Preterm birth, defined as delivery before 37 completed weeks of gestation, remains a major global public health concern and is associated with increased neonatal morbidity and mortality. Due to the immaturity of physiological systems, preterm infants are particularly vulnerable to environmental stressors such as excessive noise, bright lighting, frequent handling, and invasive medical procedures commonly encountered in neonatal intensive care units (NICUs). These stressors may lead to physiological instability, altered behavioral responses, impaired neurodevelopment, and long-term cognitive and emotional difficulties.

In addition to ensuring survival, contemporary neonatal care emphasizes supporting long-term growth, neurodevelopment, and well-being while minimizing stress and discomfort. Non-pharmacological interventions, particularly touch-based approaches, have gained prominence as safe and developmentally supportive strategies. Therapeutic Touch (TT) is a holistic nursing intervention based on the theory that the human body is surrounded by a dynamic energy field that can be balanced through intentional, gentle hand movements without invasive contact. TT has been reported to reduce pain, anxiety, and stress, while promoting relaxation and physiological stability in various patient populations.

Despite increasing interest in integrative and supportive neonatal care practices, randomized controlled trials evaluating the effects of Therapeutic Touch on preterm infants are scarce. Existing studies suggest that touch-based interventions may improve behavioral regulation, reduce stress hormone levels, support weight gain, and shorten hospital stays. However, evidence specifically addressing the impact of Therapeutic Touch on behavioral responses, comfort, and core physiological parameters in preterm infants remains limited.

This randomized controlled trial aims to systematically evaluate the effects of Therapeutic Touch administered by a trained practitioner on preterm infants hospitalized in the NICU. Outcomes will include behavioral responses, comfort levels, and physiological parameters such as heart rate, respiratory rate, oxygen saturation, and body temperature. By providing rigorous evidence on the safety and effectiveness of Therapeutic Touch in neonatal care, this study seeks to support the integration of holistic, non-pharmacological interventions into routine NICU practice and contribute to improved health and well-being outcomes for preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* Infants with a gestational age between 28-37 weeks,
* Birth weight of 1500 gr and above,
* Post-feeding,
* Hospitalized in Level 1 or Level 2 NICU,
* Stable health status will be included in the study.

Exclusion Criteria:

* Infants with:heart disease,
* congenital anomalies,
* skin health problems,
* neurological diseases,
* mechanical ventilation,
* those receiving continuous opioid, sedative, anticonvulsant or corticosteroid treatment,
* active infection or antibiotic treatment,
* undergoing surgery will be excluded from the study.

Ages: 28 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 62 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Neonatal Comfort Level | Baseline (prior to first intervention session) and Day 5 (after completion of the 5-day intervention period)
  The primary outcome of this study is the neonatal comfort level of preterm infants. Comfort will be assessed using a validated neonatal comfort scale. Measurements will be obtained at baseline and after completion of the 5-day Therapeutic Touch intervention period. Lower total scores indicate higher levels of comfort. For analysis, comfort scale scores will be compared between the Therapeutic Touch and control groups.
Behavioral Responses | Baseline (prior to first intervention session) and Day 5 (after completion of the 5-day intervention period)
  Behavioral responses of preterm infants will be assessed using a standardized neonatal behavioral assessment scale. Measurements will be obtained at baseline and after completion of the 5-day Therapeutic Touch intervention period. Lower scores indicate more positive behavioral states, while higher scores indicate negative behavioral responses. For analysis, behavioral assessment scale scores will be compared between the Therapeutic Touch and control groups.
Heart Rate | Baseline (prior to first intervention session) and Day 5 (after completion of the 5-day intervention period)
  Heart rate (beats per minute) will be measured using standard bedside monitors. Measurements will be obtained immediately before, during, and after each Therapeutic Touch session across the 5-day intervention period. For analysis, heart rate values will be summarized as mean values over the intervention period, and the post-intervention heart rate will be compared between the Therapeutic Touch and control groups.
Respiratory Rate | Baseline (prior to first intervention session) and Day 5 (after completion of the 5-day intervention period)
  Respiratory rate (breaths per minute) will be measured using standard bedside monitors. Measurements will be obtained immediately before, during, and after each Therapeutic Touch session across the 5-day intervention period. For analysis, respiratory rate values will be summarized as mean values over the intervention period, and the post-intervention respiratory rate will be compared between the Therapeutic Touch and control groups.
Oxygen Saturation | Baseline (prior to first intervention session) and Day 5 (after completion of the 5-day intervention period)
  Oxygen saturation (%) will be continuously monitored using pulse oximetry. Measurements will be obtained immediately before, during, and after each Therapeutic Touch session across the 5-day intervention period. For analysis, oxygen saturation values will be summarized as mean values over the intervention period, and post-intervention oxygen saturation levels will be compared between the Therapeutic Touch and control groups.
Blood Pressure | Baseline (prior to first intervention session) and Day 5 (after completion of the 5-day intervention period)
  Blood pressure (mmHg) will be measured using standard neonatal blood pressure monitoring methods. Measurements will be obtained immediately before, during, and after each Therapeutic Touch session across the 5-day intervention period. For analysis, blood pressure values will be summarized as mean values over the intervention period, and post-intervention blood pressure values will be compared between the Therapeutic Touch and control groups.

CONTACTS AND LOCATIONS:
Overall Officials: HABIBE BAY ÖZÇALIK, Principal Investigator — associate professor
Locations (1):
- Habibe Bay Ozcalik, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be publicly shared during the study period. After completion of the study, de-identified data may be shared with other researchers for scientific purposes upon reasonable request, in accordance with ethical regulations and institutional policies.